CLINICAL TRIAL: NCT00394706
Title: Resuscitation Outcomes Consortium (ROC) Prehospital Resuscitation Using an Impedance Valve and Early Versus Delayed Analysis
Brief Title: Resuscitation Outcomes Consortium (ROC) Prehospital Resuscitation Using an Impedance Valve
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated because preliminary data suggested no difference in the strategies.
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Defence Research and Development Canada (Industry); Heart and Stroke Foundation of Canada (Other); American Heart Association (Other)
Responsible Party: Principal Investigator, Susanne May, Principal Investigator, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 29919; HL077863
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Heart Arrest
Keywords: cardiac arrest; cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Use of Impedance Threshold Device (ITD)
  Interventions: Device: Impedance Threshold Device (ITD)
- 2 (Sham Comparator): Sham ITD
  Interventions: Device: Sham ITD
- 3 (Other): Analyze early. Upon EMS (emergency medical services) arrival at the scene of a non-traumatic cardiac arrest, the EMS providers assess the cardiac rhythm as soon as possible. Approximately thirty seconds of CPR (cardiopulmonary resuscitation) may be done prior to an assessment of the cardiac rhythm to determine whether a defibrillatory shock is required.
  Interventions: Other: Analyze early
- 4 (Other): Analyze late. Upon the EMS arrival at the scene of a non-traumatic cardiac arrest, three minutes of CPR is done prior to the assessment of the cardiac rhythm to determine whether a defibrillatory shock is required.
  Interventions: Other: Analyze later

INTERVENTIONS:
Device: Impedance Threshold Device (ITD) — Use of Impedance Threshold Device (ITD)
  Arms: 1
Device: Sham ITD — Sham ITD
  Arms: 2
Other: Analyze early — Upon EMS arrival at the scene of a non-traumatic cardiac arrest, an assessment of the cardiac rhythm is done to determine whether a defibrillatory shock is required.
  Arms: 3
Other: Analyze later — Upon EMS arrival at the scene of a non-traumatic cardiac arrest, three minutes of CPR is given prior to the assessment of the cardiac rhythm to determine whether a defibrillatory shock is required.
  Arms: 4

SUMMARY:
The purpose of this study is to look at two different treatments during a cardiac arrest that occurs outside of the hospital and whether either or both treatments will increase the number of people who live to hospital discharge. A cardiac arrest is when the heart stops pumping blood to the body.

DETAILED DESCRIPTION:
The first treatment involves using a device called the Impedance Threshold Device (ITD). The ITD is a small hard plastic device about the size of a fist that is attached to the face mask or airway tube used during CPR (cardiopulmonary resuscitation). The ITD provides increased blood flow back to the heart during chest compressions until the heart starts beating on its own again.

The other treatment involves the amount of CPR given before the emergency medical services (EMS) providers first look at the heart rhythm to determine if a shock is needed. A person would receive either about 30 seconds of chest compressions or about 3 minutes of compressions before checking the heart rhythm. Giving some compressions before checking the heart rhythm increases the blood being circulated to the body. Researchers do not know how many compressions before the rhythm check are necessary to save more lives.

Depending on the circumstances of the cardiac arrest a person may receive only one of these treatments or both of these treatments. The purpose of the research study is to determine if more people live when either the real ITD is used or if additional CPR is given before looking at the heart rhythm the first time. This study is being conducted in 9 different areas throughout the United States and Canada by the Resuscitation Outcomes Consortium (ROC). About 15,000 patients will be enrolled in this research study.

ELIGIBILITY:
Inclusion Criteria:

* All persons of local age of consent or older who suffer non-traumatic cardiopulmonary arrest outside of the hospital in the study communities with defibrillation and/or delivery of chest compressions provided by emergency medical service (EMS) providers dispatched to the scene and do not meet any of the exclusion criteria.

Exclusion Criteria:

Common:

* Do not attempt resuscitation (DNAR) orders
* Blunt, penetrating, or burn-related injury
* Patients with exsanguinations
* Known prisoners
* Known pregnancy
* Non-ROC EMS agency/provider

For Analyzing Late versus Early

* EMS-witnessed arrests
* Non-EMS rhythm analysis (AED placed by police or lay responder is an exclusion but CPR by lay or other non-EMS responders is not)

For ITD:

* Tracheostomy present
* CPR performed with the mechanical compression "Autopulse" device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11738 (Actual)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron L Weisfeldt, MD, Study Chair — Johns Hopkins University
Locations (9):
- United States (7):
  - Alabama Resuscitation Center, Birmingham, Alabama
  - UCSD-San Diego Resuscitation Center, San Diego, California
  - Portland Resuscitation Outcomes Consortium, Oregon Health & Sciences University, Portland, Oregon
  - The Pittsburgh Resuscitation Network, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Dallas Center for Resuscitation Research, University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle-King County Center for Resuscitation Research, University of Washington, Seattle, Washington
  - Milwaukee Resuscitation Network, Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Ottawa/University of British Columbia Collaborative RCC, Ottawa Health Research, Ottawa, Ontario
  - Toronto Regional Resuscitation Research Out-of-Hospital Network, University of Toronto, Toronto, Ontario

REFERENCES:
- [Background] Aufderheide TP, Nichol G, Rea TD, Brown SP, Leroux BG, Pepe PE, Kudenchuk PJ, Christenson J, Daya MR, Dorian P, Callaway CW, Idris AH, Andrusiek D, Stephens SW, Hostler D, Davis DP, Dunford JV, Pirrallo RG, Stiell IG, Clement CM, Craig A, Van Ottingham L, Schmidt TA, Wang HE, Weisfeldt ML, Ornato JP, Sopko G; Resuscitation Outcomes Consortium (ROC) Investigators. A trial of an impedance threshold device in out-of-hospital cardiac arrest. N Engl J Med. 2011 Sep 1;365(9):798-806. doi: 10.1056/NEJMoa1010821. PMID 21879897
- [Result] Stiell IG, Nichol G, Leroux BG, Rea TD, Ornato JP, Powell J, Christenson J, Callaway CW, Kudenchuk PJ, Aufderheide TP, Idris AH, Daya MR, Wang HE, Morrison LJ, Davis D, Andrusiek D, Stephens S, Cheskes S, Schmicker RH, Fowler R, Vaillancourt C, Hostler D, Zive D, Pirrallo RG, Vilke GM, Sopko G, Weisfeldt M; ROC Investigators. Early versus later rhythm analysis in patients with out-of-hospital cardiac arrest. N Engl J Med. 2011 Sep 1;365(9):787-97. doi: 10.1056/NEJMoa1010076. PMID 21879896
- [Derived] Kawano T, Grunau B, Scheuermeyer FX, Gibo K, Fordyce CB, Lin S, Stenstrom R, Schlamp R, Jenneson S, Christenson J. Intraosseous Vascular Access Is Associated With Lower Survival and Neurologic Recovery Among Patients With Out-of-Hospital Cardiac Arrest. Ann Emerg Med. 2018 May;71(5):588-596. doi: 10.1016/j.annemergmed.2017.11.015. Epub 2018 Jan 6. PMID 29310869
- [Derived] Ho ML, Gatien M, Vaillancourt C, Whitham V, Stiell IG. Utility of prehospital electrocardiogram characteristics as prognostic markers in out-of-hospital pulseless electrical activity arrests. Emerg Med J. 2018 Feb;35(2):89-95. doi: 10.1136/emermed-2017-206878. Epub 2017 Oct 21. PMID 29055890
- [Derived] Reynolds JC, Grunau BE, Rittenberger JC, Sawyer KN, Kurz MC, Callaway CW. Association Between Duration of Resuscitation and Favorable Outcome After Out-of-Hospital Cardiac Arrest: Implications for Prolonging or Terminating Resuscitation. Circulation. 2016 Dec 20;134(25):2084-2094. doi: 10.1161/CIRCULATIONAHA.116.023309. Epub 2016 Oct 19. PMID 27760796
- [Derived] Zheng R, Luo S, Liao J, Liu Z, Xu J, Zhan H, Liao X, Xiong Y, Idris A. Conversion to shockable rhythms is associated with better outcomes in out-of-hospital cardiac arrest patients with initial asystole but not in those with pulseless electrical activity. Resuscitation. 2016 Oct;107:88-93. doi: 10.1016/j.resuscitation.2016.08.008. Epub 2016 Aug 21. PMID 27554946
- [Derived] Idris AH, Guffey D, Pepe PE, Brown SP, Brooks SC, Callaway CW, Christenson J, Davis DP, Daya MR, Gray R, Kudenchuk PJ, Larsen J, Lin S, Menegazzi JJ, Sheehan K, Sopko G, Stiell I, Nichol G, Aufderheide TP; Resuscitation Outcomes Consortium Investigators. Chest compression rates and survival following out-of-hospital cardiac arrest. Crit Care Med. 2015 Apr;43(4):840-8. doi: 10.1097/CCM.0000000000000824. PMID 25565457
- [Derived] Stiell IG, Brown SP, Nichol G, Cheskes S, Vaillancourt C, Callaway CW, Morrison LJ, Christenson J, Aufderheide TP, Davis DP, Free C, Hostler D, Stouffer JA, Idris AH; Resuscitation Outcomes Consortium Investigators. What is the optimal chest compression depth during out-of-hospital cardiac arrest resuscitation of adult patients? Circulation. 2014 Nov 25;130(22):1962-70. doi: 10.1161/CIRCULATIONAHA.114.008671. Epub 2014 Sep 24. PMID 25252721
- See also: Click here for more information about the ROC PRIMED Trial — http://uwctc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical sites enrolled patients during a run-in period with the first patient enrolled on June 7, 2007. The run-in period ranged from from 2 to 6 months across the sites. The last patient was enrolled in the evaluable phase on November 6, 2009. All patients were enrolled in the pre-hospital EMS setting.
Groups:
- Analyze Early + ITD: Analyze early: upon EMS (emergency medical services) arrival at the scene of a non-traumatic cardiac arrest, the EMS providers assess the cardiac rhythm as soon as possible. Approximately thirty seconds of CPR (cardiopulmonary resuscitation) may be done prior to an assessment of the cardiac rhythm to determine whether a defibrillatory shock is required. Use of ITD (Impedance Threshold Device) by EMS providers in the prehospital setting.
- Analyze Early + Sham: Analyze early: upon EMS arrival at the scene of a non-traumatic cardiac arrest, the EMS providers assess the cardiac rhythm as soon as possible. Approximately thirty seconds of CPR may be done prior to an assessment of the cardiac rhythm to determine whether a defibrillatory shock is required. Use of a sham ITD by EMS providers in the pre-hospital setting.
- Analyze Early, Not in ITD vs Sham: Analyze early. Upon EMS arrival at the scene of a non-traumatic cardiac arrest, the EMS providers assess the cardiac rhythm as soon as possible. Approximately thirty seconds of CPR may be done prior to an assessment of the cardiac rhythm to determine whether a defibrillatory shock is required. Neither an ITD nor sham device used.
- Analyze Later + ITD: Analyze later: upon the EMS arrival at the scene of a non-traumatic cardiac arrest, three minutes of CPR is done prior to the assessment of the cardiac rhythm to determine whether a defibrillatory shock is required. Use of Impedance Threshold Device by EMS providers in the pre-hospital setting.
- Analyze Later + Sham: Analyze later: upon the EMS arrival at the scene of a non-traumatic cardiac arrest, three minutes of CPR is done prior to the assessment of the cardiac rhythm to determine whether a defibrillatory shock is required. Use of a sham ITD by EMS providers in the pre-hospital setting.
- Analyze Later, Not in ITD vs. Sham: Analyze later: upon the EMS arrival at the scene of a non-traumatic cardiac arrest, three minutes of CPR is done prior to the assessment of the cardiac rhythm to determine whether a defibrillatory shock is required. Neither an ITD nor sham device used.
- Not in AEvAL, ITD Device: Upon the EMS arrival at the scene of a non-traumatic cardiac arrest, local policy determines the length of CPR done prior to the assessment of the cardiac rhythm to determine whether a defibrillatory shock is required. Impedance Threshold Device used by EMS providers in the pre-hospital setting.
- Not in AEvAL, Sham: Upon the EMS arrival at the scene of a non-traumatic cardiac arrest, local policy determines the length of CPR done prior to the assessment of the cardiac rhythm to determine whether a defibrillatory shock is required. Sham ITD used by EMS providers in the pre-hospital setting.
Period: Overall Study
Arm/Group | Analyze Early + ITD | Analyze Early + Sham | Analyze Early, Not in ITD vs Sham | Analyze Later + ITD | Analyze Later + Sham | Analyze Later, Not in ITD vs. Sham | Not in AEvAL, ITD Device | Not in AEvAL, Sham
Started | 1819 | 1862 | 1624 | 1633 | 1636 | 1384 | 929 | 851
Completed | 1815 | 1860 | 1615 | 1632 | 1634 | 1377 | 926 | 851
Not Completed | 4 | 2 | 9 | 1 | 2 | 7 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 8 | 1 | 2 | 5 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Analyze Early + ITD | Analyze Early + Sham | Analyze Early, Not in ITD vs Sham | Analyze Later + ITD | Analyze Later + Sham | Analyze Later, Not in ITD vs. Sham | Not in AEvAL, ITD Device | Not in AEvAL, Sham | Total
Number analyzed (Participants) | 1817 | 1861 | 1621 | 1631 | 1633 | 1379 | 929 | 851 | 11722
Age, Categorical [Count of Participants; unit: Participants] — Age is not available for 8 ITD, 8 Sham, 11 Analyze Early, and 18 Analyze Later subjects.
  Participants
    <=18 years | 1 | 2 | 2 | 1 | 4 | 0 | 1 | 0 | 11
    Between 18 and 65 years | 734 | 809 | 687 | 693 | 675 | 590 | 381 | 370 | 4939
    >=65 years | 1082 | 1050 | 932 | 937 | 954 | 789 | 547 | 481 | 6772
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is not available for 8 ITD, 8 Sham, 11 Analyze Early, and 18 Analyze Later subjects.
  years | 67.3 (16.3) | 66.6 (16.4) | 66.3 (17.0) | 67.2 (16.6) | 67.1 (16.4) | 66.3 (16.7) | 67.7 (16.3) | 66.7 (16.7) | 66.9 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender missing for one ITD and one analyze earlier subject.
  Participants
    Female | 609 | 673 | 605 | 615 | 578 | 486 | 313 | 303 | 4182
    Male | 1208 | 1188 | 1016 | 1016 | 1055 | 893 | 616 | 548 | 7540
Region of Enrollment [Number; unit: participants]
  United States | 733 | 764 | 411 | 691 | 698 | 400 | 534 | 489 | 4720
  Canada | 1084 | 1097 | 1210 | 940 | 935 | 979 | 395 | 362 | 7002

OUTCOME MEASURES:

1. Primary Outcome: Survival to Hospital Discharge With Satisfactory Function (Modified Rankin Scale [MRS] of Less Than or Equal to 3).
Description: The modified Rankin Score (mRS) measures the ability of patients to function independently. The scale goes from 0 (no symptoms) to 6 (death). Subjects with a mRS scores of three or less (i.e. better) at the time of hospital discharge were considered to have a positive outcome, resulting in a binary measure.
Time Frame: Hospital discharge or death prior to discharge
Population: Analyses of both interventions excluded subjects who suffered arrest secondary to drowning, strangulation, or electrocution; or for whom the primary outcome was unknown. Additionally, the ITD vs. Sham analysis excluded subjects who did not have the device applied, had study exclusions, or who had a response time of more than 15 minutes.
Measure: Number; unit: participants
Groups:
- Analyze Early: Analyze early: upon EMS (emergency medical services) arrival at the scene of a non-traumatic cardiac arrest, the EMS providers assess the cardiac rhythm as soon as possible. Approximately thirty seconds of CPR may be done prior to an assessment of the cardiac rhythm to determine whether a defibrillatory shock is required.
- Analyze Later: Analyze later: upon the EMS arrival at the scene of a non-traumatic cardiac arrest, three minutes of CPR is done prior to the assessment of the cardiac rhythm to determine whether a defibrillatory shock is required.
- Active ITD: Use of Impedance Threshold Device by EMS providers in the pre-hospital setting.
- Sham ITD: Sham ITD used by EMS providers in the pre-hospital setting.
Arm/Group | Analyze Early | Analyze Later | Active ITD | Sham ITD
Number analyzed (Participants) | 5290 | 4643 | 4373 | 4345
participants | 310 | 273 | 254 | 260
Statistical Analysis 1: Comparison: Analyze Early vs Analyze Later; Comparison of the rates of MRS <=3 in Analyze Early vs. Analyze Later arms using a linear mixed effect model with an identity link and random effects to account for the cluster randomization; Test type: Superiority or Other; p = 0.59, Mixed Models Analysis — Two sided test with an a priori threshold of 0.05 for declaring statistical significance; Risk Difference (RD) = -0.2, 95% CI 2-sided [-1.1 to 0.7] — Estimate of the rate of MRS <= 3 in Analyze Later arm minus rate in Analyze early arm
Statistical Analysis 2: Comparison: Active ITD vs Sham ITD; Comparison of the rates of MRS <=3 in Active ITD and Sham treatment arms, adjusted for sequential monitoring; Test type: Superiority or Other; p = 0.71, t-test, 2 sided — To adjust for group sequential monitoring, the point estimate was bias-adjusted (Whitehead 1986) and confidence intervals and P values calculated from the maximum likelihood based ordering of the outcome(Emerson and Fleming, 1990); Risk Difference (RD) = -0.1, 95% CI 2-sided [-1.1 to 0.8] — Estimate of the rate of MRS <= 3 in the active ITD arm minus the rate in the Sham ITD arm

2. Secondary Outcome: Survival to Hospital Discharge
Time Frame: Survival to hospital discharge or death before discharge
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Analyze Early | Analyze Later | Active ITD | Sham ITD
Number analyzed (Participants) | 5290 | 4643 | 4373 | 4345
participants | 427 | 372 | 357 | 355
Statistical Analysis 1: Comparison: Analyze Early vs Analyze Later; Comparison of the rates of survival to hospital discharge in Analyze Early vs. Analyze Later arms using a generalized estimating equations model with an identity link, grouping on cluster; Test type: Superiority or Other; p = 0.92, GEE — Two sided test with an a priori threshold of 0.05 for declaring statistical significance; Risk Difference (RD) = -0.1, 95% CI 2-sided [-1.2 to 1.1] — Estimate of the rate of survival to hospital discharge in Analyze Later arm minus rate in Analyze early arm
Statistical Analysis 2: Comparison: Active ITD vs Sham ITD; Comparison of the rates of survival to hospital discharge in Active ITD and Sham treatment arms; Test type: Superiority or Other; p = 0.99, t-test, 2 sided; Risk Difference (RD) = 0.0, 95% CI 2-sided [-1.2 to 1.1] — Estimate of the rate of survival to hospital discharge in the active ITD arm minus rate in the Sham ITD arm

3. Secondary Outcome: Modified Rankin Score at 6 Months After Hospital Discharge
Description: The modified Rankin Score (mRS) measures the ability of patients to function independently. The scale goes from 0 (no symptoms) to 6 (death).
Time Frame: 6 months post hospital discharge
Population: ITT population, survived to hospital discharge, consented to participate in the post-discharge substudy, and with at least one post-discharge assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Analyze Early | Analyze Later | Active ITD | Sham ITD
Number analyzed (Participants) | 308 | 274 | 218 | 223
units on a scale | 1.7 (1.8) | 1.8 (1.8) | 1.8 (1.9) | 1.6 (1.7)
Statistical Analysis 1: Comparison: Analyze Early vs Analyze Later; Linear regression was used to assess associations between post-discharge measures and treatment group comparisons with adjustment for baseline characteristics. Site was adjusted for to accommodate clustering of patients within sites. All regression analyses used robust standard errors to accommodate non-constant variances; Test type: Superiority; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.20 to 0.34] — Mean MRS for Analyze Later minus mean MRS for Analyze Early (i.e. positive values favor Analyze Later)
Statistical Analysis 2: Comparison: Active ITD vs Sham ITD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.17 to 0.44] — Mean MRS for Active ITD minus mean MRS for Sham ITD (i.e. positive values favor the active device)

4. Secondary Outcome: Adult Lifestyle and Function Version of Mini-Mental Status Exam at 6 Months
Description: The adult lifestyle and function interview (ALFI) version of the mini-mental status exam (MMSE) measures neurological status. The ALFI-MMSE has 23 items. It is scored from 0 to 22, with lower scores interpreted as being worse.
Time Frame: 6 months post hospital discharge
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Analyze Early | Analyze Later | Active ITD | Sham ITD
Number analyzed (Participants) | 318 | 265 | 214 | 226
units on a scale | 18.3 (6.0) | 18.5 (5.5) | 18.0 (6.3) | 18.7 (5.5)
Statistical Analysis 1: Comparison: Analyze Early vs Analyze Later; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.71 to 0.83] — Mean ALFI-MMSE for Analyze Later minus mean ALFI-MMSE for Analyze Early (i.e. positive values favor Analyze Later)
Statistical Analysis 2: Comparison: Active ITD vs Sham ITD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.61 to 0.28] — Mean ALFI-MMSE for Active ITD minus mean ALFI-MMSE for Sham ITD (i.e. positive values favor the active device)

5. Secondary Outcome: Health Utilities Index III Score and Geriatric Depression Scale Score 6 Months
Description: The Health Utilities Index Mark 3 system was used to evaluate generic health related quality of life (HRQL). The interview-administered version of HUI3 requires completion of a maximum of 39 questions. The HUI3 consists of eight attributes of general health (vision, hearing, speech, mobility, dexterity, emotion, cognition, and pain) with five or six levels per attribute. For each respondent, health status is described as a vector that combines the levels of each attribute. This information is then converted into a utility score of HRQL on a scale from perfect health (1.0) to death (0).
Time Frame: 6 months post hospital discharge
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Analyze Early | Analyze Later | Active ITD | Sham ITD
Number analyzed (Participants) | 273 | 240 | 191 | 189
units on a scale | 0.74 (0.34) | 0.73 (0.35) | 0.71 (0.36) | 0.75 (0.33)
Statistical Analysis 1: Comparison: Analyze Early vs Analyze Later; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.06 to 0.05] — Mean HUI for Analyze Later minus mean HUI for Analyze Early (i.e. positive values favor Analyze Later)
Statistical Analysis 2: Comparison: Active ITD vs Sham ITD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.08 to 0.05] — Mean HUI for Active ITD minus mean HUI for Sham ITD (i.e. positive values favor the active device)

ADVERSE EVENTS:
Arm/Group | Analyze Early + ITD | Analyze Early + Sham | Analyze Early, Not in ITD vs Sham | Analyze Later + ITD | Analyze Later + Sham | Analyze Later, Not in ITD vs. Sham | Not in AEvAL, ITD Device | Not in AEvAL, Sham
Serious Adverse Events (participants affected / at risk) | 154/2310 | 193/2321 | 122/2051 | 166/2156 | 174/2191 | 121/1839 | 181/1336 | 152/1278
Other Adverse Events (participants affected / at risk) | 0/2310 | 0/2321 | 0/2051 | 0/2156 | 0/2191 | 0/1839 | 0/1336 | 0/1278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Analyze Early + ITD (N=2310) | Analyze Early + Sham (N=2321) | Analyze Early, Not in ITD vs Sham (N=2051) | Analyze Later + ITD (N=2156) | Analyze Later + Sham (N=2191) | Analyze Later, Not in ITD vs. Sham (N=1839) | Not in AEvAL, ITD Device (N=1336) | Not in AEvAL, Sham (N=1278)
Airway bleeding (Respiratory, thoracic and mediastinal disorders) | 62 (64) | 79 (79) | 28 (28) | 67 (67) | 67 (69) | 26 (28) | 60 (61) | 51 (51) — Finding of frank blood or bloody fluids in the airway secretions, the oro- or naso-pharynx region, or the advanced airway by EMS or ED/hospital personnel.
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 98 (99) | 120 (121) | 98 (98) | 104 (104) | 118 (118) | 99 (101) | 134 (135) | 108 (109)
Defibrillator burns to chest (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver lacerations (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Liver lacerations secondary to CPR with bleeding and hypotension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes